CLINICAL TRIAL: NCT00562055
Title: Phase 2, Randomized, Double-Blind, Parallel-Group, Four Week, Efficacy And Safety Trial Of [S,S]-Reboxetine (PNU-165442g) And Atomoxetine In Adults With Attention Deficit Hyperactivity Disorder.
Brief Title: Double-Blind, Four Week Trial Of [S,S]-Reboxetine And Atomoxetine In Adults With Attention Deficit Hyperactivity Disorder.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was withdrawn due to business reasons.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6061060; A6061060
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: PNU-165442G; [S,S]-reboxetine
- Arm B (Active Comparator)
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine
  Arms: Arm B
Drug: PNU-165442G; [S,S]-reboxetine
  Arms: Arm A

SUMMARY:
This study will compare the safety and efficacy of [S,S]-reboxetine to atomoxetine in the treatment of adult patients with attention deficity-hyperactivity disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Attention Deficit Hyperactivity Disorder according to DSM-IV criteria.
2. Score of 24 or higher on the Adult ADHD Investigator Symptom Rating Scale
3. Score of 4 or higher on the Clinician Global Impression - Severity scale

Exclusion Criteria:

1. Significant comorbid psychiatric diagnoses
2. Significant risk of suicidal or violent behavior

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11

PRIMARY OUTCOMES:
Adult ADHD Investigator Symptom Rating Scale - Total Score | 4 weeks

SECONDARY OUTCOMES:
Adult ADHD Investigator Symptom Rating Scale - Inattention Subscale Score | 4 weeks
Adult ADHD Investigator Symptom Rating Scale - Hyperactivity/Impulsivity Subscale Score | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061060&StudyName=DOUBLE-BLIND%2C%20FOUR%20WEEK%20TRIAL%20OF%20%5BS%2CS%5D-REBOXETINE%20AND%20ATOMOXETINE%20IN%20ADULTS%20WITH%20ATTENTION%20DEFICIT%20HYPERACTIVITY%20DISORDER